CLINICAL TRIAL: NCT05312580
Title: A Retrospective PMCF Study Evaluating the Safety and Clinical Performance of the S.M.A.R.T. Flex Stent Iliac, S.M.A.R.T. Flex SFA/PP, S.M.A.R.T. Control Nitinol Stent, S.M.A.R.T. Nitinol Stent, PALMAZ Blue .018 Peripheral Stent on Slalom, PALMAZ Genesis .035 Peripheral Stent on Opta Pro, SABER OTW PTA Catheter, SABERX PTA Dilatation Catheter and PowerFlex Pro PTA Catheter for the Endovascular Interventions in the Ilio-femoropopliteal Vessels
Brief Title: PMCF Study for Peripheral Arteries Above the Knee (ATK)
Status: Completed | Type: Observational
Sponsor: Cordis US Corp. (Industry)
Collaborators: FCRE (Foundation for Cardiovascular Research and Education) (Other)
Responsible Party: Sponsor
Other Study IDs: FCRE-220105_ATK
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Arterial Disease; Femoropopliteal Stenosis; Angiopathy, Peripheral
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The rationale of this study is to confirm and support the clinical safety and performance of the products in a real-word population of 350 patients who underwent an endovascular intervention within standard-of-care (SOC) of the ilio-femoropopliteal artery, using at least 1 of the products (named above) from Cordis US Corp.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is >18 years old at conduction of the procedure.
2. Patient who underwent endovascular procedure of the ilio-femoropopliteal vessel with at least one of the following the S.M.A.R.T. Flex Stent Iliac and/or S.M.A.R.T. Flex SFA/PP and/or S.M.A.R.T. Control Nitinol Stent and/or S.M.A.R.T. Nitinol Stent and/or PALMAZ Blue .018 Peripheral Stent on Slalom and/or PALMAZ Genesis .035 Peripheral Stent on Opta Pro and/or SABER OTW PTA Catheter and/or SABERX PTA Dilatation Catheter and/or PowerFlex Pro PTA Catheter as described in the IFU of the devices.
3. Target Lesion is located in the ilio-femoropopliteal vessels.

Exclusion Criteria:

1. Anatomy or size of vessels that did not allow appropriate usage of the devices, following IFU of the devices.
2. Known contraindication and/or allergy to (a component of) the device as described in the IFU of the devices.
3. Women who were pregnant or lactating at the time of the procedure.
4. Life expectancy of less than 12 months at the time of procedure.
5. Any patient who was hemodynamically unstable at onset of procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who underwent endovascular procedure of the ilio-femoropopliteal vessel with at least one of the above mentioned study devices.
Sampling Method: Non-Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Freedom from Serious Adverse Events | 30 days
  Acute primary Safety Endpoint:
  Freedom from Serious Adverse Events (SAEs) and Serious Adverse Device Effect (SADEs) during the procedure and up to 30 days after the procedure.
Freedom from Serious Adverse Events | 12 months
  Primary Safety Endpoint:
  Freedom from Serious Adverse Events (SAEs) and Serious Adverse Device Effect (SADEs) up to 12 months after the procedure.
Technical success rate | During the procedure
  Acute Primary Efficacy Endpoint:
  Technical success rate defined as successful crossing, introduction, deployment (stents)/deflation (balloon catheter) and a <30% residual stenosis on visual assessment of S.M.A.R.T. Flex Stent Iliac, S.M.A.R.T. Flex SFA/PP, S.M.A.R.T. Control Nitinol Stent, S.M.A.R.T. Nitinol Stent, PALMAZ Blue .018 Peripheral Stent on Slalom, PALMAZ Genesis .035 Peripheral Stent on Opta Pro, SABER OTW PTA Catheter, SABERX PTA Dilatation Catheter and PowerFlex Pro PTA Catheter according to the respective IFU.
Freedom from clinically-driven target lesion revascularization | 12 months
  Primary Efficacy Endpoint:
  The primary efficacy endpoint is freedom from clinically-driven target lesion revascularization (CD-TLR) at 12 months, defined as any reintervention at the target lesion due to symptoms.

SECONDARY OUTCOMES:
Technical success rate | During the procedure
  Technical success rate defined as successful crossing, introduction, deployment and successful completion of the procedure of the Cordis guidewires (Emerald, ATW, Stablizer, Storq, SV 0.018", Wizdom) and/or the Cordis guiding catheters (Adroit, Vista Brite Tip) and/or the Cordis diagnostic catheters (Super Torque, Super Torque MB, Super Torque Plus, Infiniti 4F/5F/6F, Tempo 4F, Tempo Aqua, High Flow, Pigtail Straightener) and/or the Cordis vascular access devices (Avanti+, Brite Tip, Vista Brite IG, vessel dilator) and/or the Cordis vascular closure devices (MynxGrip and Mynx Control) and/or the Cordis OUTBACK CTO catheters according to the respective IFU.
Technical success rate | Day of procedure
  Technical success rate defined as successful hemostasis without conversion to manual/mechanical compression of the Cordis vascular closure devices (MynxGrip and Mynx Control) according to the respective IFU.
Freedom from CD-TLR | 36- and 60-months
  Freedom from clinically-driven target lesion revascularization (CD-TLR) at 36- and 60-months, defined as any reintervention at the target lesion due to symptoms.
Stent fracture rate | Up to 30 days post-procedure, 12-, 36- and 60-months
  Stent fracture rate assessed at up to 30 days post-procedure, 12-, 36- and 60-months.
Stent migration rate | Up to 30 days post-procedure, 12-, 36- and 60-months
  Stent migration rate assessed at up to 30 days post-procedure, 12-, 36- and 60-months.
Change of Ankle Brachial Index | Up to 30 days post-procedure, 12-, 36- and 60-months
  Change of Ankle Brachial Index (ABI) assessed at up to 30 days post-procedure, 12-, 36- and 60-months compared to baseline ABI.
Time-to-hemostasis | Day of procedure
  Time-to-hemostasis assessed for the Cordis vascular closure devices (MynxGrip and Mynx Control). Categorized as Hemostatic time category (HTC) ≤2, HTC >2 to ≤4, HTC >4 to ≤5, HTC >5 to ≤7, HTC >7 to ≤10 min.
Time-to-ambulation | Day of procedure
  Time-to-ambulation assessed for the Cordis vascular closure devices (MynxGrip and Mynx Control) defined as time between end of the procedure and ambulation in hours.
Rate of Major Amputation free survival | Up to 30 days post-procedure, 12-, 36- and 60-months
  Rate of Major Amputation free survival defined as any amputation above the knee assessed at up to 30 days post-procedure, 12-, 36- and 60-months.
Clinical success | Up to 30 days post-procedure, 12-, 36- and 60-months
  Clinical success at up to 30 days post procedure, 12-, 36- and 60-months, defined as an improvement of the Rutherford Classification of one class or more, as compared to the pre-procedure Rutherford Classification.
Vessel perforation/dissection | During the procedure
  Vessel perforation/dissection during the procedure.
Freedom from Serious Adverse Events (SAEs) and Serious Adverse Device Events (SADEs) | 36- and 60-months
  Freedom from Serious Adverse Events (SAEs) and Serious Adverse Device Events (SADEs) at 36- and 60-months after the procedure.
All cause of mortality | procedure through study completion (12 months)
  All cause of mortality through life of the study.

CONTACTS AND LOCATIONS:
Locations (9):
- Austria (4):
  - Medizinische Universität Innsbruck, Innsbruck
  - KABEG-Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Universitätsklinikum St. Pölten - Lilienfeld, Sankt Pölten
  - Medizinische Universität WienMedizinische Universität Wien, Vienna
- France (4):
  - Public health establishment, Arras Hospital, Arras
  - Hospital de la Timone, Marseille
  - The Public Hospital, Centre Hospitalier Universitaire de Toulouse, Toulouse
  - Clinique River Gauche, Toulouse
- Leiden University Medical Center (LUMC), Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No